CLINICAL TRIAL: NCT00169091
Title: Clozapine or Haloperidol in First Episode Schizophrenia
Brief Title: Clozapine Versus Haloperidol for Treating the First Episode of Schizophrenia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Dartmouth-Hitchcock Medical Center (Other); Commonwealth Research Center, Massachusetts (Other); Novartis (Industry)
Responsible Party: Principal Investigator, AlanGreen, Chair, Department of Psychiatry Geisel School of Medicine at Dartmouth, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH052376 (NIH); R01MH052376 (NIH)
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Schizophrenia
Keywords: Clozapine; Haloperidol; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Clozapine; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Clozapine (Experimental): Clozapine 12.5-300 mg taken orally per day for 12 weeks in the acute phase of the study and up to 130 weeks (total) in the Follow-up portion of the study.
  Interventions: Drug: Clozapine
- Haloperidol (Active Comparator): Haloperidol 2-12 mg taken orally per day for 12 weeks in the acute phase of the study and up to 130 weeks (total) in the Follow-up portion of the study.
  Interventions: Drug: Haloperidol

INTERVENTIONS:
Drug: Clozapine — Medication will be divided into twice daily dosing and administered in a blinded fashion. The medication will be tapered from 12.5 mg on Day 1 to up to 300 mg on Day 12.
  Other Names: Clozaril
  Arms: Clozapine
Drug: Haloperidol — Medication will be divided into twice daily dosing and administered in a blinded fashion. The medication will be tapered from 2 mg on Day 1 to up to 12 mg on Day 12.
  Other Names: Haldol
  Arms: Haloperidol

SUMMARY:
This study will examine the physical responses brought on by clozapine and haloperidol in people experiencing their first episode of schizophrenia.

DETAILED DESCRIPTION:
This is a longitudinal double blind, 2- 5 year study of the clinical, neuroendocrine and biochemical response to clozapine (CLOZ) and haloperidol (HAL) in a group of "first episode" schizophrenic (RDC) patients. Within the protocol, we compare the differential effects of the two drugs over the short term (12 weeks) and the long-term (2-5 years); we evaluate the relationship between change in prolactin level and clinical response of the patients; and we search for biochemical predictors and correlates of clinical response. To achieve the study aims, we employ a drug-washout period, a 12-week acute treatment period; and an 88 - 260 week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* RDC diagnosis of schizophrenia
* Men and women, without regard to race/ethnicity,
* Aged 18-45
* Acutely psychotic with a score of at least 3 on one of the psychotic scale items of the Brief Psychiatric Rating Scale (BPRS) (hallucinations, delusions, conceptual disorganization) and a total BPRS of > 21 (on a 0 - 6 scale);
* Require treatment with neuroleptic drugs on a clinical basis;
* The patient (or the patient's authorized legal representative) must understand the nature of the study and sign the informed consent;
* Be within the first episode of a psychotic disorder;
* Have a history of neuroleptic treatment of < 12 weeks;
* Likely to remain in the study for 2 years.

Exclusion Criteria:

* Substance dependence in the last six months
* History of seizure or blood dyscrasia
* Major medical illness
* Pregnancy or Lactation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 1996-03; Primary Completion 2003-09 (Actual); Study Completion 2003-10

PRIMARY OUTCOMES:
Brief Psychiatric Rating Scale | Weekly during the Acute Treatment Phase and every two weeks in Follow-Up
  This study will use the 24 item BPRS

CONTACTS AND LOCATIONS:
Overall Officials: Alan I Green, MD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- Commonwealth Research Center, Jamaica Plain, Massachusetts, United States

REFERENCES:
- [Background] Green AI, Schildkraut JJ. Should clozapine be a first-line treatment for schizophrenia? The rationale for a double-blind clinical trial in first-episode patients. Harv Rev Psychiatry. 1995 May-Jun;3(1):1-9. doi: 10.3109/10673229509017159. PMID 9384923